CLINICAL TRIAL: NCT01955291
Title: The Role of Virtual Therapy by Means of Reinforced Feedback in Virtual Environment on Upper Limb Function in Post-stroke Patients.
Brief Title: Reinforced Feedback in Virtual Environment
Acronym: RFVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Camillo, Venezia, Italy (Other)
Responsible Party: Principal Investigator, Pawel Kiper, PhD, IRCCS San Camillo, Venezia, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02/09 vers. 2.0
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Stroke
Keywords: Virtual Reality, Motor Learning, Rehabilitation, Upper Limb
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reinforced Feedback in Virtual Environment (Experimental): During the experiment, patients in the RFVE training group (Reinforced Feedback in Virtual Environment) will receive 1 hour of virtual reality-based therapy by means of RFVE and 1 hour of TNR treatment (Traditional Neuromotor Rehabilitation). Both treatments will last 1 hour a day, five days weekly for four weeks. The treatment is focused on motor function impairment of the upper extremity.
  Interventions: Device: Reinforced Feedback in Virtual Environment (RFVE)
- Traditional Neromotor Rehabilitation (Other): The TNR training group (Traditional Neuromotor Rehabilitation) patients will be treated totally for two hours daily by means of a TNR programme. The treatment will last 4 weeks.
  Interventions: Other: Traditional Neuromotor Rehabilitation

INTERVENTIONS:
Device: Reinforced Feedback in Virtual Environment (RFVE) — The patients allocated to RFVE group, will be treated using the "Virtual Reality Rehabilitation System" (VRRS). During the virtual therapy the subject will be seated in front of the wall screen grasping a sensorized real object with the affected hand. If the grasp is not possible the sensors will be fixed on a glove worn by the patient. The real object held by the subject, equipped with electromagnetic sensors, is matched to the virtual handling object. Thereafter, the patient moved the real object (e.g. ball) following the trajectory of the corresponding virtual object displayed on the computer screen in accordance with the requested virtual task.
  Other Names: Virtual Reality Rehabilitation System (VRRS)
  Arms: Reinforced Feedback in Virtual Environment
Other: Traditional Neuromotor Rehabilitation — The patients randomized to the Traditional Neuromotor Rehabilitation group will be asked to perform exercises for postural control, exercises for hand pre-configuration, exercises for the stimulation of manipulation and functional skills, exercises for proximal-distal coordination. All the exercises will be performed with or without the assistance of a physiotherapist. The upper limb motricity will be trained with progressive complexity. To achieve the requested goal (in a horizontal or vertical plane) patients will be asked to perform various movements, for example: shoulder flexion and extension, shoulder abduction and adduction, shoulder internal and external rotation and shoulder circumduction, elbow flexion and extension, forearm pronation and supination, hand grasping-release and clenching into a fist.
  Arms: Traditional Neromotor Rehabilitation

SUMMARY:
The aims of the study is to explore whether the rehabilitation of the upper extremity performed in interaction with a virtual environment could improve motor function in post-ischemic and post-haemorrhagic stroke subjects with hemiparesis, in comparison to the traditional neuromotor rehabilitation treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients affected by a stroke occurring in the period no longer than 1 year before the enrolment
* both first ischemic and hemorrhagic stroke
* subjects who did not had RFVE treatment previously
* scoring higher than 24 points in the Mini-Mental State Examination test

Exclusion Criteria:

* upper extremity complete hemiplegia
* upper limbs sensory disorders
* clinical evidence of cognitive impairment
* neglect
* apraxia
* comprehension difficulties
* post-traumatic injury of the upper limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2008-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Fugl_Meyer Upper Extremity scale (F-M UE) | 20 min
  Applied at the beginning and at the end of treatment 4 weeks thereafter.

SECONDARY OUTCOMES:
Functional Independence Measure scale (FIM) | 20 min
  Assessed at the beginning and at the end of treatment 4 weeks thereafter.
National Institutes of Health Stroke Scale (NIHSS) | 5 min
  Assessed at the beginning and at the end of treatment 4 weeks thereafter.
Kinematic assessment | 30 min
  The kinematic assessment include the execution of standardised upper limb movements, such as: forearm pronation and supination, elbow flexion and extension, shoulder abduction and adduction, shoulder internal and external rotation, shoulder flexion and extension and reaching movements. The mean linear velocity (Speed), the mean duration of movements (Time) and the mean number of submovements (Peak) will be measured, by means of the Virtual Reality Rehabilitation System (VRRS). The data will be registered at the beginning and at the end of treatment, 4 weeks thereafter.

OTHER OUTCOMES:
Edmonton Symptom Assessment Scale (ESAS) | 5 min
  Assessed at the beginning and at the end of the treatment, 4 weeks thereafter.
Modified Ashworth scale | 10 min
  Assessed at the beginning and at the end of the treatment, 4 weeks thereafter. The scale consist of evaluation of 5 muscles; pectoralis major, biceps, wrist flexors, flexor digitorum superficialis, flexor digitorum profundus.
Mini Mental State Examination scale (MMSE) | 20 min
  Performed at the beginning.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Tonin, MD, Study Director — Fondazione Ospedale San Camillo IRCCS
Locations (1):
- Fondazione Ospedale San Camillo IRCCS, Venezia, Veneto, Italy

REFERENCES:
- [Background] Laver K, George S, Thomas S, Deutsch JE, Crotty M. Cochrane review: virtual reality for stroke rehabilitation. Eur J Phys Rehabil Med. 2012 Sep;48(3):523-30. Epub 2012 Jun 20. PMID 22713539
- [Background] Kiper P, Agostini M, Luque-Moreno C, Tonin P, Turolla A. Reinforced feedback in virtual environment for rehabilitation of upper extremity dysfunction after stroke: preliminary data from a randomized controlled trial. Biomed Res Int. 2014;2014:752128. doi: 10.1155/2014/752128. Epub 2014 Mar 13. PMID 24745024
- [Derived] Kiper P, Szczudlik A, Agostini M, Opara J, Nowobilski R, Ventura L, Tonin P, Turolla A. Virtual Reality for Upper Limb Rehabilitation in Subacute and Chronic Stroke: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2018 May;99(5):834-842.e4. doi: 10.1016/j.apmr.2018.01.023. Epub 2018 Feb 14. PMID 29453980